CLINICAL TRIAL: NCT03650010
Title: Evaluation of Epidemiology and Radiological and Clinical Outcomes in Total Ankle Prosthesis
Brief Title: Total Ankle Replacement: Clinical and Radiological Outcomes
Status: Recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Principal Investigator, Elena Cittera, FEDERICO USUELLI, MD PRINCIPAL INVESTIGATOR, I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio
Other Study IDs: Tarus
Record Dates: First submitted 2017-12-08; First posted 2018-08-28 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Ankle Arthritis
MeSH Terms: interventions — Arthroplasty, Replacement, Ankle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Procedure: Total ankle replacement — total ankle prosthesis through a lateral or an anterior approach

SUMMARY:
This retrospective and prospective study intends to evaluate the epidemiology and effectiveness of ankle joint surgery in patients operated from January 2011 to March 2026, evaluating the results both clinically and radiographically.

DETAILED DESCRIPTION:
The aim of this study is to evaluate radiographically and clinically using clinical and radiographic outcomes . Few studies exist in the literature and rarely report fix-bearing and mobile-bearing prosthetics [1-4]. Therefore the data related to this study can be considered a reference in the literature.

Patients who performed and will perform ankle prosthesis surgery from January 2011 to March 2026 and who underwent a clinical evaluation (also using questionnaires and scores) and radiographic evaluation.

The clinical data and radiological parameters were collected together with the visits and the procedures prescribed according to the clinical routine of the department.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* age ≥ 18 years at the time of surgery
* patients who underwent ankle replacement surgery from January 2011 to March 2026

Exclusion Criteria:

- age < 18 years at the time of surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1066 patients who underwent total ankle replacement
Sampling Method: Probability Sample
Enrollment: 1066 (Estimated)
Dates: Start 2016-05-11 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Changes in American orthopaedic foot and ankle society (AOFAS) ankle-hindfoot score | Pre operatively, 2 months post-operatively, 6 months post-operatively, 12 months post-operatively, 24-36-48-60-72-84-96-108-120 months post-operatively
  The American orthopaedic foot and ankle society (AOFAS) ankle-hindfoot score combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient (to assess sagittal motion, hindfoot motion, ankle-hindfoot stability and alignment of the ankle-hindfoot). The scale includes nine items that can be divided into three subscales (pain, function and alignment). Pain consists of one item with a maximal score of 40 points, indicating no pain. Function consists of seven items with a maximal score of 50 points, indicating full function. Alignment consists of one item with a maximal score of 10 points, indicating good alignment. The maximal score is 100 points, indicating no symptoms or impairments.
Changes in Short form 12 (SF 12) | Pre operatively, 2 months post-operatively, 6 months post-operatively, 12 months post-operatively, 24-36-48-60-72-84-96-108-120 months post-operatively
  The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey (Ware, Kosinski, and Keller, 1996). The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life. Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Anterior distal tibial angle | Pre operatively
  (ADTA: normal value 83.0 ± 3.6 degrees). The angle is subtended by the anatomic axis of the tibia and the line connecting the distal points on the anterior and posterior tibial articular surface on the anterior side (Figure 1). The tibia axis was defined as the line connecting the centres of two circles designed over the proximal and the distal tibia adjusting their radius to the anterior and posterior tibial cortices.
Changes in beta angle | 2 months post-operatively, 6 months post-operatively, 12 months post-operatively, 24-36-48-60-72-84-96-108-120 months post-operatively
  β-angle (normal value 85.0 ± 2.0 degrees). This angle is subtended anteriorly by the longitudinal axis of the tibia and the articular surface of the tibial component on the lateral view
Changes in alpha angle | 2 months post-operatively, 6 months post-operatively, 12 months post-operatively, 24-36-48-60-72-84-96-108-120 months post-operatively
  the α-angle is formed by the angle between the anatomic axis of the tibia and the articular surface of the tibial component on the AP view (normal value 90.0 ± 2.0 degrees)
Medial distal tibial angle | Pre operatively
  It is the angle between the anatomic axis of the tibia and the line connecting the distal point on the medial and lateral articular surface. (normal value 92.4 ± 3.1 degrees).

SECONDARY OUTCOMES:
Changes in visual analogue scale | Pre operatively, 2 months post-operatively, 6 months post-operatively, 12 months post-operatively, 24-36-48-60-72-84-96-108-120 months post-operatively
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale. When responding to a VAS item, respondents specify their level of agreement to a statement by indicating a position along a continuous line between two end-points.

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Galeazzi, Milan, Milano, Italy

IPD SHARING:
Plan to Share IPD: Undecided